CLINICAL TRIAL: NCT01784523
Title: A Prospective Randomized Controlled Trial of Hydroxychloroquine in the Primary Thrombosis Prophylaxis of aPL Positive But Thrombosis-free Patients.
Brief Title: Hydroxychloroquine for the First Thrombosis Prevention in Antiphospholipid Antibody Positive Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low recruitment rate exacerbated by manufacturing shortage and price increase of hydroxychloroquine.
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: AntiPhospholipid Syndrome Alliance For Clinical Trials and InternatiOnal Networking (Unknown); The New York Community Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014-253; NCT02635126 (obsolete NCT alias)
Record Dates: First submitted 2013-02-03; First posted 2013-02-06 (Estimated); Results first posted 2021-05-04 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-08

CONDITIONS: Antiphospholipid Syndrome
Keywords: antiphospholipid autoantibodies; antiphospholipid positive
MeSH Terms: conditions — Antiphospholipid Syndrome | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard treatment (No Intervention): patients randomized to standard treatment will not receive hydroxychloroquine.
- Hydroxychloroquine (Experimental): Patients will be randomized to receive standard of care or standard of care + hydroxychloroquine. Dose will be weight-adjusted: 200 mg daily for patients weighing <60kg; and 400 mg daily (200 mg twice a day)for patients weighing >60kg.
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine
  Other Names: plaquenil
  Arms: Hydroxychloroquine

SUMMARY:
In this multi-center international study, our aim is to determine the effectiveness of HCQ for primary thrombosis prophylaxis in persistently aPL-positive but thrombosis-free patients without systemic autoimmune diseases.

DETAILED DESCRIPTION:
Randomized to receive HCQ or no treatment in addition to their standard regimen. 11 study visits and 10 phone visits over 5 years.

This study was terminated at 2 years due to low recruitment rate exacerbated by manufacturing shortage and price increase of hydroxychloroquine.

ELIGIBILITY:
Inclusion Criteria:

* Persistent(at least 12 weeks apart)aPL-positivity within 12 months prior to the screening defined as:

  * aCL IgG/M (>40U,medium-to-high titer,and/or greater than the 99th percentile)and/or
  * aβ2GPI IgG/M(>40U, medium-to-high titer, and/or greater than the 99th percentile)and/or
  * Positive LA test based on the International Society of Thrombosis & Haematosis Recommendations

Selected Exclusion Criteria:

* History of thrombosis (arterial, venous, and/or biopsy proven microthrombosis
* History of Transient Ischemic Attack Confirmed by a Neurologist
* SLE Diagnosis based on the ACR Classification Criteria > 4/11
* Other Systemic Autoimmune Diseases diagnosed based on ACR Classification Criteria
* Current Hydroxychloroquine or another antimalarial treatment (-3 months)
* Current warfarin treatment (-3 months)
* Current heparin therapy( -3 months)
* Current pregnancy
* History of Hydroxychloroquine eye toxicity
* History of Hydroxychloroquine allergy
* Known glucose-6-phosphate dehydrogenase deficiency

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2013-02; Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doruk Erkan, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Erkan D, Lockshin MD; APS ACTION members. APS ACTION--AntiPhospholipid Syndrome Alliance For Clinical Trials and InternatiOnal Networking. Lupus. 2012 Jun;21(7):695-8. doi: 10.1177/0961203312437810. PMID 22635205
- [Background] Erkan D, Derksen R, Levy R, Machin S, Ortel T, Pierangeli S, Roubey R, Lockshin M. Antiphospholipid Syndrome Clinical Research Task Force report. Lupus. 2011 Feb;20(2):219-24. doi: 10.1177/0961203310395053. PMID 21303838
- See also: APS ACTION — http://www.apsaction.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydroxychloroquine: Patients will be randomized to receive standard of care or standard of care + hydroxychloroquine. Dose will be weight-adjusted: 200 mg daily for patients weighing <60kg; and 400 mg daily (200 mg twice a day)for patients weighing >60kg.
  Hydroxychloroquine
Period: Overall Study
Arm/Group | Standard Treatment | Hydroxychloroquine
Started | 7 | 4
Completed | 0 | 0
Not Completed | 7 | 4
Not completed — Study closed early | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment | Hydroxychloroquine | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (8.98) | 45.75 (7.89) | 44.64 (8.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Acute Thrombosis Event
Description: To determine the efficacy of Hydroxychloroquine in the primary thrombosis prevention of persistently aPL-positive but thrombosis free patients with no other systemic autoimmune diseases over the five year study period.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment | Hydroxychloroquine
Number analyzed (Participants) | 7 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Standard Treatment | Hydroxychloroquine
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4
Other Adverse Events (participants affected / at risk) | 0/7 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No